CLINICAL TRIAL: NCT01898156
Title: Two-Part, Open-Label, Multi-Center, Phase 1/2 Study of Anti-GM2 Ganglioside Monoclonal Antibody BIW-8962 as Monotherapy in Subjects With Previously Treated Advanced/Recurrent Lung Cancer or Mesothelioma
Brief Title: Two-Part, Open-Label, Multi-Center, Phase 1/2 Study of BIW-8962 as Monotherapy in Subjects With Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8962-002
Record Dates: First submitted 2013-06-18; First posted 2013-07-12 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Phase 1 Portion : Non Small Cell Lung Cancer(NSCLC), Small Cell Lung Cancer(SCLC), Mesothelioma; Phase 2 Portion : Small Cell Lung Cancer(SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Mesothelioma | interventions — BIW-8962

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIW-8962 (Experimental): Phase 1 - Dose escalation based on the BIW-8962 tolerability and safety data obtained from three subjects enrolled in a cohort (first cycle of treatment), enrollment at the next dose level or additional subjects into the ongoing cohort will occur
  Phase 2 - Recommended dose determined in Phase 1
  Interventions: Drug: BIW-8962

INTERVENTIONS:
Drug: BIW-8962 — Phase 1 -With a standard 3+3 dose escalation design, the enrollment in Phase 1 will proceed until the MTD has been defined or the highest dose level has been reached. BIW-8962 will be administered intravenously on day 1 of each 21 day cycle.
  Phase 2 - RP2D of BIW-8962 determined in phase 1 portion will be administered until progression or unacceptable toxicity develops.

SUMMARY:
This Phase 1/2 study is designed to assess the following: safety and tolerability of BIW-8962, Dose Limiting Toxicities (DLTs), Maximum Tolerated Dose (MTD), Recommended Phase 2 Dose (RP2D) in Phase 1 in subjects with advanced/recurrent lung cancers or mesothelioma and preliminary efficacy in Phase 2 in subjects with advanced/recurrent Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: histopathological-documented, measurable or non-measurable unresectable, advanced primary or recurrent SCLC, NSCLC or mesothelioma
* Phase 2: measurable, unresectable advanced or recurrent SCLC
* A life expectancy > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1 at study entry
* Echocardiogram or multigated acquisition (MUGA) scan with left ventricular ejection fraction (LVEF) ≥ 50%, or ≥ institution's established lower limit of normal
* Adequate hematologic, hepatic, renal and lung function

Exclusion Criteria:

* Subject received cytotoxic anti-cancer chemotherapy, orally available signaling pathway-targeted therapy, hormonal therapy, radiotherapy, immunotherapy, or investigational agents within 3 weeks prior to the first dose
* Subject received monoclonal antibodies within 4 weeks of the first dose
* Major surgery within 4 weeks prior to the first dose
* Known symptomatic brain metastases
* Clinically significant cardiovascular disease
* Leptomeningeal disease
* Uncontrolled intercurrent illness including ongoing or active infection, uncontrolled diabetes, etc
* Known HIV disease or acquired immunodeficiency syndrome-related illness
* A psychiatric illness, disability or social situation
* Hypersensitivity reaction to monoclonal antibodies, other therapeutic proteins
* A history of primary brain/CNS malignancy
* Neurological paraneoplastic syndrome

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Phase 1 - To determine Maximum Tolerated Dose(MTD) | First 3-week cycle of treatment
  Phase 1 -Adverse Event collection and assessment will be done for all potentially treated subjects to assess the safety, tolerability, and determine the DLTs, maximum tolerated dose (MTD).
Phase 2 - To assess the objective response rate(Partial Response and Complete Response) | Until Progressive Disease (PD) determined
  Phase 2 - Tumor response and progression will be evaluated every 6 weeks using RECIST v 1.1. Partial Response (PR) or Complete Response (CR) will be confirmed 4 weeks after first detection of response.

SECONDARY OUTCOMES:
Phase 1 - To evaluate preliminary efficacy | Until Progressive Disease (PD) determined
  Phase 1 - Tumor response progression will be evaluated using RECIST V1.1 for the assessment of efficacy
Phase 1 - To determine the q3w pharmacokinetic profile of BIW-8962 | Pre-dose, and Day 1, 2, 3, 5, 8, 12 and 15 in Cycle 1 and 3, Pre-dose in Cycle 2, 4, 5,and up to Cycle 6
  Phase 1 - Pharmacokinetic (PK) parameters such as Maximum concentration (Cmax), time to maximum concentration (Tmax), minimum concentration(Cmin), area under the curve (AUC), half-life (t1/2), clearance (CL), and etc., are assessed.
Phase 2 - To assess safety and tolerance | Every 3 weeks, until 45days after the last dose or within 7 days prior to the initiation of subsequent anti-cancer treatment
  Phase 2 - All safety information will be collected and then evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin Korea, Seoul, South Korea